CLINICAL TRIAL: NCT01747486
Title: Dose Optimization Trial of Autologous T Cells Engineered to Express Anti-CD19 Chimeric Antigen Receptor (CART-19) in Patients With Relapsed or Refractory CD19+ Chronic Lymphocytic Leukemia (CLL)
Brief Title: Dose Optimization Trial of CD19 Redirected Autologous T Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 03712, 816556
Record Dates: First submitted 2012-12-10; First posted 2012-12-11 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2019-08

CONDITIONS: Adult Patients Who Have Relapsed or Refractory CLL (3rd Line) or SLL
MeSH Terms: interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Target dose of 1-5x10e8 (Experimental): Arm 1: Target dose of 1-5x10e8 CART-19 cells (calculated as range of 10-50% transduced cells in 1 x10e9 total cells)
  Interventions: Biological: CART-19
- Target dose of 1-5x10e7 (Experimental): Arm 2: Target dose of 1-5x10e7 CART-19 cells (calculated as the range of 10-50% transduced cells in 1 x10e8 total cells)
  Interventions: Biological: CART-19

INTERVENTIONS:
Biological: CART-19 — CART-19 cells (autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCR zeta and 4-1BB costimulatory domains)

SUMMARY:
This is a randomized, open-label, parallel group study to determine the optimal dose of CART-19 cells (autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCR Zeta and 4-1 BB co-stimulatory domains) of the two dose levels being assessed (1-5x10e8 vs. 1-5x10e7 CART-19 cells). This trial will be conducted in two stages.

DETAILED DESCRIPTION:
This study is being conducted to determine the optimal dose of autologous CART-19 T cells engineered to express anti-CD19 chimeric antigen receptors in patients with relapsed or refractory CD19 positive chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL). The two dose levels being assessed are 1-5x10e8 versus 1-5x10e7. The trial will be conducted in two stages. In stage I subjects will be randomized into one of the two dose cohort with a1:1 ratio for a total of 12 subjects per dose cohort. Stage II will be to enroll an additional 8 subjects to the selected dose cohort once safety, tolerability and clinical responses have been evaluated to determine the optimal dose cohort.

ELIGIBILITY:
Inclusion Criteria

* Documented CD19+ CLL or SLL
* Successful test expansion of T-cells
* At least 2 prior chemotherapy regimens, not including single agent monoclonal antibody (rituxan) therapy. Single agent ofatumumab will be counted as a regimen. -Patients with high risk disease manifested by deletion chromosome 17p will be eligible if they fail to achieve a CR to initial therapy or progress within 2 years of 1 prior regimen.
* Patients who progress within 2 years after the second or higher line of therapy will be eligible. For instance, patients who had progression < 2 years after second or greater line therapy, but who have responded to their most recent treatment (3rd line or higher) will be eligible.
* Subject is not appropriate candidate for a potentially curative allogeneic SCT due to the state of disease, co-morbid illness, lack of an available donor, or patient declines Performance status (ECOG) 0 or 1
* Age >/= 18 years
* Adequate organ system function including:

  1. Creatinine < 1.6 mg/dl
  2. ALT/AST < 3x upper limit of normal
  3. Total Bilirubin <2.0 mg/dl
* Any relapse after prior autologous SCT will make patient eligible regardless of other prior therapy
* Patients with relapsed disease after prior allogeneic SCT (myeloablative or nonmyeloablative) will be eligible if they meet all other inclusion criteria and:

  1. Have no active GVHD and require no immunosuppression
  2. Are more than 6 months from transplant
* No contraindications for leukapheresis
* Left Ventricular Ejection fraction >40%
* Gives voluntary informed consent

Retreatment Inclusion Criteria

* Performance Status 0-1
* Adequate organ system function including:

  * Creatinine < 1.6 mg/dl
  * ALT/AST < 3x upper limit of normal
  * Total Bilirubin < 2.0 mg/dl
* Subject is not an appropriate candidate for a potentially curative allogeneic SCT due to the state of disease, co-morbid illness, lack of an available donor, or patient declines.
* Left Ventricular Ejection Fraction > 40%
* No contraindications for leukapheresis (if required for retreatment)
* Gives voluntary informed consent for retreatment

Exclusion Criteria

* Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion.
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. For additional details regarding use of steroid and immunosuppressant medications.
* Any uncontrolled active medical disorder that would preclude participation as outlined
* HIV infection
* Patients with active CNS involvement with malignancy. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment.
* Class III/IV cardiovascular disability according to the New York Heart Association Classification

Retreatment Exclusion Criteria

* Pregnant or lactating women. Female study participants must have a negative serum or urine pregnancy test performed within 48 hours before infusion.
* Uncontrolled active infection
* Active hepatitis or hepatitis infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* HIV infection
* Patients with active CNS involvement with malignancy. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment on the retreatment cohort.
* Class III/IV cardiovascular disability according to the New York Heart Association Classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2018-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramsonc Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] van Bruggen JAC, Martens AWJ, Fraietta JA, Hofland T, Tonino SH, Eldering E, Levin MD, Siska PJ, Endstra S, Rathmell JC, June CH, Porter DL, Melenhorst JJ, Kater AP, van der Windt GJW. Chronic lymphocytic leukemia cells impair mitochondrial fitness in CD8+ T cells and impede CAR T-cell efficacy. Blood. 2019 Jul 4;134(1):44-58. doi: 10.1182/blood.2018885863. Epub 2019 May 10. PMID 31076448
- [Derived] Fraietta JA, Beckwith KA, Patel PR, Ruella M, Zheng Z, Barrett DM, Lacey SF, Melenhorst JJ, McGettigan SE, Cook DR, Zhang C, Xu J, Do P, Hulitt J, Kudchodkar SB, Cogdill AP, Gill S, Porter DL, Woyach JA, Long M, Johnson AJ, Maddocks K, Muthusamy N, Levine BL, June CH, Byrd JC, Maus MV. Ibrutinib enhances chimeric antigen receptor T-cell engraftment and efficacy in leukemia. Blood. 2016 Mar 3;127(9):1117-27. doi: 10.1182/blood-2015-11-679134. Epub 2016 Jan 26. PMID 26813675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Enrolled - 02-Jan-2013 Last Patient Completed - 13-Dec-2017
Pre-assignment Details: Study was conducted in 2 stages. Stage 1: subjects were randomized into one of the two arms (Arm 1: Higher dose & Arm 2 : Lower dose) Stage 2: the selected dose cohort was expanded to enroll additional subjects. Based on the Stage 1 analysis performed in Nov 2014, Arm 1 was chosen for expansion in Stage 2 and enrolled additional 12 subjects.
Period: Stage 1
Arm/Group | Target Dose of 1-5x10e8 | Target Dose of 1-5x10e7
Started | 15 | 15
Completed | 3 | 2
Not Completed | 12 | 13
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Disease progression | 4 | 9
Not completed — Death | 1 | 1
Period: Stage 2
Arm/Group | Target Dose of 1-5x10e8 | Target Dose of 1-5x10e7
Started | 12 | 0
Completed | 3 | 0
Not Completed | 9 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — New Cancer Therapy | 3 | 0
Not completed — Disease Progression | 3 | 0

BASELINE CHARACTERISTICS:
Population: In high dose cohort, 15 patients were enrolled in Stage 1 and 12 were in stage 2.
Groups:
- Target Dose of 1-5x10e8: Arm 1: Target dose of 1-5x10e8 CART-19 cells (calculated as range of 10-50% transduced cells in 1 x10e9 total cells)
  CART-19: CART-19 cells (autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCR zeta and 4-1BB costimulatory domains)
  Note: For baseline measures, subjects from stage 1 (15) and stage 2 (12) are combined to have total 27 subjects. In stage 2, higher dose arm (arm 1) was chosen based on the stage 1 analysis performed to expand and enrolled 12 additional subjects.
- Target Dose of 1-5x10e7: Arm 2: Target dose of 1-5x10e7 CART-19 cells (calculated as the range of 10-50% transduced cells in 1 x10e8 total cells)
  CART-19: CART-19 cells (autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCR zeta and 4-1BB costimulatory domains)
  Note: In stage 1, 15 subject were enrolled in this arm. Since this arm was not chosen for stage 2, no additional subjects were enrolled. total subjects in this arm were 15.
- Total: Total of all reporting groups
Arm/Group | Target Dose of 1-5x10e8 | Target Dose of 1-5x10e7 | Total
Number analyzed (Participants) | 27 | 15 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 12 | 31
  >=65 years | 8 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 21 | 11 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 26 | 15 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 15 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Complete Response Within 3 Months
Description: Complete response (including complete response with incomplete marrow recovery) within 3 months (in evaluable patients). The eveluable set comprise of patients who have received CART19 at intended dose level and completed at least 3-month follow-up after the infusion or discontinued due to disease progression, new cancer therapy or death.
Time Frame: 3 months
Population: The Evaluable Set comprised all patients who received high dose (1-5×10^8) or low dose (1-5×10^7) CTL019 transduced cells as randomized, and completed at least 3-month follow-up after the infusion or discontinued due to disease progression, new cancer therapy or death.
Measure: Count of Participants; unit: Participants
Arm/Group | Target Dose of 1-5x10e8 | Target Dose of 1-5x10e7
Number analyzed (Participants) | 18 | 13
Participants
  Complete Response (CR) | 1 | 1
  CR with incomplete marrow recovery (CRi) | 5 | 0
  Partial Response (PR) | 4 | 2
  PR with incomplete marrow recovery (PRi) | 0 | 1
  No Response (NR)/ Progressive Disease (PD) | 8 | 9

ADVERSE EVENTS:
Time Frame: For this study, adverse events were collected until the subject is off study or until the end of study visit at 12 months before subjects were enrolled into separate long term follow up study.
Groups:
- Target Dose of 1-5x10e8: Arm 1: Target dose of 1-5x10e8 CART-19 cells (calculated as range of 10-50% transduced cells in 1 x10e9 total cells)
  CART-19: CART-19 cells (autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCR zeta and 4-1BB costimulatory domains)
  Note: For this group, subjects from stage 1 (15) and stage 2 (12) are combined to have total 27 subjects. In stage 2, higher dose arm (arm 1) was chosen based on the stage 1 analysis performed to expand and enrolled 12 additional subjects.
Arm/Group | Target Dose of 1-5x10e8 | Target Dose of 1-5x10e7
All-Cause Mortality (participants affected / at risk) | 6/27 | 6/15
Serious Adverse Events (participants affected / at risk) | 23/27 | 9/15
Other Adverse Events (participants affected / at risk) | 24/27 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Target Dose of 1-5x10e8 (N=27) | Target Dose of 1-5x10e7 (N=15)
Cytokine Release Syndrome (Immune system disorders) | 12 | 6
Pyrexia (General disorders) | 5 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 4
Pneumonia (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Acute kideny injury (Renal and urinary disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Target Dose of 1-5x10e8 (N=27) | Target Dose of 1-5x10e7 (N=15)
White blood cell count decreased (Investigations) | 8 | 9
Anaemia (Blood and lymphatic system disorders) | 12 | 7
Fatigue (General disorders) | 10 | 6
CD4 lymphocytes decreased (Investigations) | 10 | 11
Pyrexia (General disorders) | 4 | 8
Cytokine release syndrome (Immune system disorders) | 12 | 6
Lymphocyte count decreased (Investigations) | 8 | 4
Nausea (Gastrointestinal disorders) | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 5
Chills (General disorders) | 3 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 4
Neutropenia (Blood and lymphatic system disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 3 | 3
Neutrophil count decreased (Investigations) | 6 | 6
Hypotension (Vascular disorders) | 2 | 4
Oedema peripheral (General disorders) | 2 | 4
Platelet count decreased (Investigations) | 5 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Post procedural infection (Infections and infestations) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0
Aspratate aminotransferase increased (Investigations) | 3 | 0
Headche (Nervous system disorders) | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT01747486/Prot_SAP_001.pdf